CLINICAL TRIAL: NCT06500169
Title: Golf Recreational Exercise for Enhanced Survivorship in Prostate Cancer Survivors Undergoing Hormone Therapy (GREENS)
Brief Title: Golf Recreational Exercise for Enhanced Survivorship in Prostate Cancer Survivors
Acronym: GREENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4P-23-4; NCI-2023-09213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-23-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-05-24; First posted 2024-07-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Localized Prostate Carcinoma; Locally Advanced Prostate Carcinoma; Stage I Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Interviews as Topic; Restraint, Physical; Exercise Test; Recreation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (golf program) (Experimental): Patients participate in the golf training program composed of group sessions over 1-2 hours with a PGA professional two times per week for ten weeks. Training consists of complimentary/warm up exercises integrated with pelvic floor muscle training, golf instruction, golf practice, and golf play on a Par 3 public golf course. Patients also wear an activity tracker and undergo blood sample collection on the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Discussion; Other: Exercise Intervention; Other: Interview; Other: Medical Device Usage and Evaluation; Procedure: Physical Examination; Other: Physical Performance Testing; Other: Questionnaire Administration; Other: Recreational Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Discussion — Ancillary studies
  Other Names: Discuss
Other: Exercise Intervention — Complete golf related exercises
Other: Interview — Ancillary studies
Other: Medical Device Usage and Evaluation — Wear activity tracker
Procedure: Physical Examination — Ancillary studies
  Other Names: Assessment; General Examination; Physical; Physical Assessment; Physical Exam; Physical examination procedure (procedure); physical_exam
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies
Other: Recreational Therapy — Participate in golf program

SUMMARY:
This clinical trial evaluates a golf recreational exercise program for enhancing survivorship in underrepresented prostate cancer survivors. Golf is a multimodal recreational activity that requires participants to utilize all muscle groups to perform the golf swing, walk over hilly and uneven terrain, maintain balance during putting and squat-like tasks. Physical activity and exercise are beneficial to physical function, cognitive function, psychosocial health, and overall quality of life during prostate cancer survivorship. These aspects of health are impacted by prostate cancer treatment, especially androgen deprivation therapy. Additionally, supervised, group-based activity programs facilitate participation in physical activity. Researchers want to examine the changes in functional abilities, psychosocial health, and quality of life following participation in in a golf program designed for prostate cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To recruit, screen, and enroll prostate cancer survivors. II. To examine the safety, feasibility, and adherence, of the 10-week (wk) GREENS program.

III. To analyze the pre-post intervention data and examine the effects (assessed by Hedges g) of the program on:

IIIa. Physical capacity; IIIb. Psychosocial wellness; IIIc. Health, and; IIId. Cognition.

OUTLINE:

Patients participate in the golf training program composed of group sessions over 1-2 hours with a Professional Golfers' Association of America (PGA) professional two times per week for ten weeks. Training consists of complimentary/warm up exercises integrated with pelvic floor muscle training, golf instruction, golf practice, and golf play on a Par 3 public golf course. Patients also wear an activity tracker and undergo blood sample collection on the study.

After completion of study intervention, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* First time, primary diagnosis of prostate cancer (PCa)
* Currently receiving androgen deprivation therapy (ADT) and/or androgen receptor blocker) for more than 6 months
* Older adult male: 55-85 years old
* The ability to stand independently without external support
* No or minimal golf experience (played < 5 times in the past 10 years)
* English speaking

Exclusion Criteria:

* Second cancer diagnosis (excluding non-invasive skin cancers) or bone metastases
* Prostatectomy less than 6 months prior to study enrollment (prostatectomy is not a requirement for study entry)
* Symptomatic cardiovascular disease, active angina, uncontrolled hypertension (systolic blood pressure (SBP) > 160 or diastolic blood pressure (DBP) > 90, high resting pulse heart rate (HR) > 90), symptomatic orthostatic hypotension
* Unstable asthma, exacerbated chronic obstructive pulmonary disease (COPD]
* History of injury or orthopedic operation within the last 6 months
* Movement disorders (e.g., Parkinson's disease (PD) or other neurological disorders), hemiparesis or paraparesis
* Severe vision or hearing problems

Ages: 55 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Up to 3 years
  Will be defined as the final number of enrolled individuals / the number of qualified individuals screened.
Participant adherence to the program | Up to 3 years
  Will be assessed by the number of participants who adhere to the study and attend > 80% of supervised training sessions.
Cost of the program | Up to 3 years
  Will be assessed by the cost that the program will be < $1,000/participant.
Staff adherence | Up to 3 years
  Will be assessed by trained staff who attend > 90% of scheduled sessions.
Program accommodations | Up to 3 years
  Will be defined as the program accommodating course scheduling for > 95% of training sessions.
Incidence of adverse events | Up to 3 years
  Will be assessed across all participants, and defined by less than 3 program-related adverse events (AEs) and any/all AEs will be mild (grade 3 or below according to Common Terminology Criteria for Adverse Events version 5).
Quality of life scores | Up to 3 years
  Will be assessed by the Functional Assessment of Cancer Therapy - Prostate (FACT-P), a 39-item self-reported questionnaire. FACT-P scores range from 0 to 156, with higher scores indicating a better quality of life. It is expected that the scores will improve with medium to large effect sizes and exceed the established minimal clinically important difference (MCID).
Circulating inflammatory biomarker levels | Up to 3 years
  Will be assessed by C-reactive protein and tumor necrosis factor alpha (TNFa) which are indicators of inflammation. Based on prior study, C-reactive protein and TNFa levels are expected to decrease with medium to large effect sizes and exceed the calculated MCID levels.
Senior fitness test scores | Up to 3 years
  Will be assessed by Short physical performance battery (SPPB). The SPPB is scored out of 12 points and higher score indicates better performance. The SPPB is a reliable (intraclass correlation coefficient [ICC] was between 0.82-0.92) and validated (MDC=2; MCID=1-3) measure for physical capacity in community-dwelling and clinical older adults.
Gait speed | Up to 3 years
  Will be assessed with self-selected gait and fast gait using a 10-feet designated walkway and timing device. Faster gait speeds in both condition indicate higher physical capacity. For reference, men in the 60-65 years age group, gait speeds over 1.53 m/s is considered above 80th percentile.
Balance Confidence | Up to 3 years
  Will be assessed by Activities-specific Balance Confidence (ABC) scale, a 16-item self-reported questionnaire. The ABC is scored from 0% to 100%, where higher scores indicate greater confidence in maintaining balance during activities.
Cognitive function | Up to 3 years
  Will be assessed by the Food and Drug Administration approved Sway Medical application (app) designed to assess cognition with a smart phone device and will be used to assess cognitive function. The app includes validated tests for processing speed, sensory processing, neuromotor response speed, inhibition, memory, and executive function, which are areas of cognitive function that are potentially influenced by prostate cancer treatments. The app has established normative values for different age group and will be used as reference.
Participant feedback of the program | Up to 3 years
  Will be assessed by a semi-structured focus group that will be conducted post intervention where participants will be asked about positive affect and negative affect associated with the intervention, their perceived mastery of different components of golf (i.e. putting, chipping, golf swing, etiquette, rules, etc.), facilitators and barriers that pertained to their participation in the intervention. These assessments will provide information unique to prostate cancer survivors and be used directly to improve the protocol and intervention design for future studies in this population. The facilitators and barriers will also be compared to established ones reported by Sattar et al. to qualitatively assess whether they are similar with our diverse cohort of minority participants located in Los Angeles, California.

CONTACTS AND LOCATIONS:
Overall Officials: George Salem, PhD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California